CLINICAL TRIAL: NCT04750252
Title: An Open Label Study to Evaluate Safety and Tolerability of StroMel™ in Subjects with Moderate to Severe Osteoarthritis of the Knee Joint
Brief Title: Safety and Tolerability of StroMel™ in Subjects with Moderate to Severe Osteoarthritis of the Knee Joint
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akan Biosciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StroMel-01
Record Dates: First submitted 2021-02-08; First posted 2021-02-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Osteo Arthritis Knee
Keywords: Stem cell, MSC, autologous, adipose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with moderate to severe OA of the Knee (Experimental)
  Interventions: Biological: StroMel

INTERVENTIONS:
Biological: StroMel — Autologous MSC

SUMMARY:
The aim of this trial is to evaluate the safety and tolerability of autologous StroMel™ for the treatment of moderate to severe OA of the knee joint.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between the ages of 25-65 years
2. Body Mass Index (BMI) less than 40 kg/m2
3. Ambulatory and in good general health as described by vital signs (blood pressure 90/60 mm Hg to 120/80 mm Hg, pulse rate 60-100 beats per minute, temperature 97.2-99.1 °F) and normal blood chemistry.
4. Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain score of ≥ 11 (worst possible = 20) over the previous 7 days
5. OA of the knee with Kellgren and Lawrence radiographic classification (Grade 2-4 inclusive) within the last 6 months
6. Minimum score of 40 out of possible 100 on the VAS (Visual Analog Scale) for pain.
7. Patients who have failed to adequately respond for at least 6 months to at least 2 OA therapies that include conservative, non-pharmacological therapy and simple analgesics (e.g., acetaminophen); nonsteroidal anti-inflammatory drugs (NSAIDS); avoidance of activities that cause joint pain; exercise; weight loss; physical therapy; and removal of excess fluid from the knee.
8. Have suitable knee joint anatomy for intra-articular injection.
9. For adults of reproductive potential: use of effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

Exclusion Criteria:

1. Reactive arthritis, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease.
2. Subject with an infection that requires parenteral antibiotic administration.
3. Active infection or crystal disease in the index joint within 1 month of screening
4. History of fracture in the index limb, joint instability, or history of acute dislocation within 12 months of screening, or fracture with sequelae at any time
5. Intra-articular treatment of any joint with any of the following agents within 6 months of screening: Any corticosteroid preparation (investigational or marketed), sodium hyaluronate, any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection); investigational six months prior to enrollment.
6. Presence of surgical hardware or other foreign body in the index joint
7. Subjects who were administered with immunosuppressants such as cyclosporin A or azathioprine within 6 weeks before screening.
8. Planned or anticipated surgery of the joint during the study period
9. Allergies to anesthesia
10. Subjects who tested positive for HIV, HCV, WNV, CMV, HBV, HTLV, ZIKA, syphilis, flu or COVID-19. Note: CMV is not a relevant communicable disease agent. A subject who tests positive or reactive for CMV is not necessarily ineligible. Physicians will determine donor eligibility for subjects with positive CMV test results.
11. History of lipid disorders: lipedema, lipomatosis, or lipodystrophies.
12. Active cancer, chemotherapy, or other malignancies in the last 6 months.
13. Recent history of DVT or pulmonary embolism requiring anticoagulants or other medicines per the hematologist.
14. Subject who participated in another clinical trial within 3 months before the screening visit
15. Any illness which, in the Investigator's judgment, will interfere with the subject's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results.
16. Subjects who are breastfeeding
17. Subjects with uncontrolled arrhythmias
18. Subjects with hemophilia; factor II, V, VII, X, or XII deficiencies; or Von Willebrand's disease.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety of StroMel in subjects with moderate to severe OA of the kneee | 12 months
  Presence of adverse events in less than 10% of the study population. Adverse events assessed will be Grade 4 administrative site infection, Grade 3 hypersensitivity/anaphylaxis, >20% increase in WOMAC pain score, treatment-related disability, and presence of tumors post-treatment.
Overall Safety of StroMel | 12 months
  Summary of all study related AEs and SAEs.

SECONDARY OUTCOMES:
Efficacy of StroMel in managing OA of the knee | 52 weeks
  Reduction of NSAIDS, until study completion
Efficacy of StroMel in assessment of OA of the knee post-treatment | 52 weeks
  Percent change from baseline in rating scales (WOMAC and VAS assessments)

CONTACTS AND LOCATIONS:
Locations (1):
- Mukesh, Gaithersburg, Maryland, United States

IPD SHARING:
Plan to Share IPD: No